CLINICAL TRIAL: NCT00484952
Title: Multicenter Study for Surveillance of Hospitalizations Due to Rotavirus-Associated Diarrhea and Estimation of the Economic Burden of Rotavirus Hospitalizations
Brief Title: Surveillance of Hospitalizations Due to Rotavirus Infections Among Children From Israel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Tel Aviv University (Other); Laniado Hospital (Other); Carmel Medical Center (Other); The Meshulash Research and Development Center Kfar Qaraa (Unknown); Ministry of Health, Israel (Other Government)
Other Study IDs: 48/2006
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-06

CONDITIONS: Rotavirus Infections
Keywords: rotavirus; diarrheal diseases; hospitalizations; multicenter; children; under five year old; Hospitalization due to diarhheal diseases; Hospitalization due to rotavirus gastroenteritis; Nosocomial rotavirus infections
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives

1. To determine the burden and characteristics of rotavirus-associated hospitalizations among children under five years of age of northern Israel
2. To identify potential risk factors of rotavirus infections associated with hospitalizations among Jewish and Arab children younger than five years of age.

Methods:

Study design: A two-year prospective study and a nested case control study will be carried out Collection of data: Questionnaires will be filled in with demographic characteristics of patients and data on the clinical manifestation of the diarrheal episode leading to hospitalization. Stool specimens will be systematically collected from all children hospitalized because of diarrheal diseases and examined for rotavirus and for bacterial and protozoan enteropathogens. Positive samples for rotavirus will be tested for G and P genotypes.

For the nested case control study additional data will be obtained from parents' interviews on variables such as: parents' education, parents' age, parents' occupation, no. of siblings, age of siblings, breastfeeding etc. to identify potential risk factors for rotavirus diarrhea necessitating hospitalization.

Data analysis: Methods of descriptive statistics / epidemiology will be applied to determine the characteristics of the burden of rotavirus-associated hospitalizations (the distribution of diarrhea associated hospitalizations by etiology, rates of rotavirus diarrheal diseases in Jewish and Arab children, age specific rates of rotavirus infections, the percentage of hospitalizations due to rotavirus diarrhea by month, etc.

For the nested case control study, univariate analysis will be first performed using Student t test for continuous variables and chi square test for categorical variables to study the statistical significance of predictive factors of rotavirus diarrheal diseases necessitating hospitalization. Multivariate analysis using logistic regression models will be performed to study the independent effect of each variable. Odds ratios (OR) and 95% CI will be computed for each variable. Two tailed p < 0.05 will be considered significant.

DETAILED DESCRIPTION:
Rationale: Vaccination against rotavirus is the most appropriate mean for prevention and control of rotavirus infections. Israel is highly endemic for diarrheal diseases but limited data exist on the burden & epidemiology of rotavirus diarrheal diseases. Such data are essential to assess the relevance of potential future vaccination against rotavirus-associated gastroenteritis in Israel.

Objectives

1. To determine the burden and characteristics of rotavirus-associated hospitalizations among children under five years of age of northern Israel
2. To identify potential risk factors of rotavirus infections associated with hospitalizations among Jewish and Arab children younger than five years of age.

Methods:

Study design: A two-year prospective study and a nested case control study will be carried out Study population: About 45000 children aged less than five years, residing in the catchment areas of three pediatric wards of sentinel hospitals (Laniado - Netanya, Carmel - Haifa & Hillel Yaffe -Hadera) will be under daily surveillance for hospitalizations due to rotavirus diarrheal diseases for two years. The catchment area of the 3 hospitals has a good representation of both Jewish and Arab pediatric population. During the study period we expect 400 hospitalizations due to diarrheal diseases and 80 hospitalizations due to rotavirus gastroenteritis annually, in each of the three hospitals (i.e. 480 cases of rotavirus- diarrheal disease in the two year study). 100 subjects hospitalized because of rotavirus associated diarrhea and 100 controls matched by age, gender and origin will be recruited for the nested case-control study.

Collection of data: Questionnaires will be filled in with demographic characteristics of patients and data on the clinical manifestation of the diarrheal episode leading to hospitalization. Stool specimens will be systematically collected from all children hospitalized because of diarrheal diseases and examined for rotavirus and for bacterial and protozoan enteropathogens. Positive samples for rotavirus will be tested for G and P genotypes.

For the nested case control study additional data will be obtained from parents' interviews on variables such as: parents' education, parents' age, parents' occupation, no. of siblings, age of siblings, breastfeeding etc. to identify potential risk factors for rotavirus diarrhea necessitating hospitalization.

Data analysis: Methods of descriptive statistics / epidemiology will be applied to determine the characteristics of the burden of rotavirus-associated hospitalizations (the distribution of diarrhea associated hospitalizations by etiology, rates of rotavirus diarrheal diseases in Jewish and Arab children, age specific rates of rotavirus infections, the percentage of hospitalizations due to rotavirus diarrhea by month, etc.

For the nested case control study, univariate analysis will be first performed using Student t test for continuous variables and chi square test for categorical variables to study the statistical significance of predictive factors of rotavirus diarrheal diseases necessitating hospitalization. Multivariate analysis using logistic regression models will be performed to study the independent effect of each variable. Odds ratios (OR) and 95% CI will be computed for each variable. Two tailed p < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age: under five year old
* Hospitalization due diarrheal disease within the study period in the pediatric wards participating in the study
* Controls: hospitalization due non-gastrointestinal causes within the study period in the pediatric wards participating in the study

Exclusion Criteria:

* Refusal

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2007-09; Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dani Cohen, PhD, Principal Investigator — Tel Aviv University
Locations (2):
- Israel (2):
  - Carmenl Medical Center, Haifa
  - Laniado Medical Center, Netanya